CLINICAL TRIAL: NCT07278336
Title: A Phase 1 First-in-Human, Open-Label Study Evaluating Safety, Pharmacokinetics, and Efficacy of ABBV-901 as a Monotherapy and in Combination With Bevacizumab in Adult Subjects With Ovarian Cancer
Brief Title: A Study to Assess Adverse Events, Change in Disease Activity and How Intravenous (IV) ABBV901 Moves Through the Body Alone or in Combination With Bevacizumab in Adult Participants With Ovarian Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M25-760; 2025-522209-40 (Other: EU CT)
Record Dates: First submitted 2025-12-02; First posted 2025-12-12 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Epithelial Ovarian, Fallopian Tube, and Primary Peritoneal Cancers; ABBV-901; Bevacizumab
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Part 1: ABBV-901 Dose Escalation (Experimental): Participants will receive escalating doses of ABBV-901 alone, as part of the approximately 3 year study duration.
  Interventions: Drug: ABBV-901
- Part 2: ABBV-901 Optimization/Expansion Dose A (Experimental): Participants will receive ABBV-901 dose A alone, as part of the approximately 3 year study duration.
  Interventions: Drug: ABBV-901
- Part 2: ABBV-901 Optimization/Expansion Dose B (Experimental): Participants will receive ABBV-901 dose B alone, as part of the approximately 3 year study duration.
  Interventions: Drug: ABBV-901
- Part 2: ABBV-901 Optimization/Expansion Dose C (Experimental): Participants will receive ABBV-901 dose C alone, as part of the approximately 3 year study duration.
  Interventions: Drug: ABBV-901
- Part 3: ABBV-901 + Bevacizumab Escalation (Experimental): Participants will receive escalating doses of ABBV-901 in combination Bevacizumab, as part of the approximately 3 year study duration.
  Interventions: Drug: ABBV-901; Drug: Bevacizumab
- Part 4: ABBV-901 + Bevacizumab Expansion (Experimental): Participants will receive the recommended doses for expansion doses of ABBV-901 in combination Bevacizumab, as part of the approximately 3 year study duration.
  Interventions: Drug: ABBV-901; Drug: Bevacizumab

INTERVENTIONS:
Drug: ABBV-901 — Intravenous (IV)
Drug: Bevacizumab — IV
  Arms: Part 3: ABBV-901 + Bevacizumab Escalation; Part 4: ABBV-901 + Bevacizumab Expansion

SUMMARY:
Ovarian cancer (OC) is a lethal disease. The purpose of this study is to assess the safety, pharmacokinetics and efficacy of ABBV901, alone or in combination with bevacizumab, in participants with ovarian cancer.

ABBV901 is an investigational drug for the treatment of ovarian cancer. This study has 4 Parts (Arms) where participants will receive ABBV-901, alone or in combination with the standard available therapy, bevacizumab. Around 207 participants will be enrolled in the study at approximately 75 sites around the world.

In part 1, participants will receive escalating doses of intravenous (IV) ABBV-901 alone. In part 2, participants will receive 1 of 3 doses of IV ABBV-901, alone to determine the optimized dose. In part 3, participants will receive escalating doses of IV ABBV-901, combination with IV bevacizumab. In part 4, participants will receive recommended doses for expansion of IV ABBV-901, combination with IV bevacizumab. The total study duration will be approximately 3 years.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic and may require frequent medical assessments, blood tests, and scans.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of an advanced or unresectable malignant high grade serous epithelial ovarian, fallopian tube, and primary peritoneal cancers (EOC), fallopian tube or primary peritoneal cancer by histology (World Health Organization [WHO] criteria).
* Participants must be considered platinum resistant. Platinum resistant disease is defined as radiographic progression within 6 months (up to 182 days) after the last dose of the most recent platinum therapy).
* Prior anticancer therapy:

  * Must have received appropriate standard of care therapy and be appropriate for participation in a Phase I study in the opinion of the investigator.
  * Platinum-resistant, high grade serous EOC cannot have had more than 5 prior lines of therapy, with clinical progression of disease on no more than 2 prior therapies since the development of platinum resistance.
* For participants enrolled in backfill, subjects must provide consent to paired biopsies which are pretreatment and on-treatment tumor biopsies from the same tumor lesion.

Exclusion Criteria:

* Ovarian Cancer (OC) with histologies other than high grade serous OC including endometrioid, low grade, clear cell, mucinous, or borderline ovarian tumor.
* Prior therapy with an antibody-drug conjugate containing a topoisomerase inhibitor.
* Prior history of Grade >= 2 ILD or pneumonitis.
* History of interstitial lung disease (ILD) or pneumonitis that required treatment with systemic steroids, nor any evidence of active ILD or pneumonitis on Screening chest computed tomography (CT) scan.
* Must not have systemically used known strong cytochrome P450 (CYP)3A inhibitors or inducers within 14 days or 5 half-lives of the drug (whichever is shorter) prior to the first dose of the study drug through the end of the DLT observation period. If clinically indicated, strong CYP3A inhibitors and inducers may be used with caution after the dose-limiting toxicity (DLT) period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Estimated)
Dates: Start 2025-11-27 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AE) | Up to Approximately 3 Years
  An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product, and which does not necessarily have a causal relationship with this treatment.
Overall Response | Up to Approximately 3 Years
  Overall response is defined as participants achieving confirmed complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 as assessed by the investigator.

SECONDARY OUTCOMES:
Duration of Response (DOR) | Up to Approximately 3 Years
  DOR is defined for participants achieving a confirmed PR or better as the time from the initial response of PR (or better) per investigator review according to RECIST Version 1.1 criteria to disease progression or death of any cause, whichever occurs earlier.
Progression-free survival (PFS) | Up to Approximately 3 Years
  PFS is defined as time from first study treatment to a documented disease progression according to RECIST Version 1.1 (or other assessment criteria), as determined by the investigator, or death due to any cause, whichever occurs earlier.
Overall Survival (OS) | Up to Approximately 3 Years
  OS is defined as time from first study treatment to death due to any cause.
Disease Control Rate | Up to Approximately 3 Years
  Disease Control Rate is defined as the percentage of participants with best overall response (BOR) of stable disease (SD), PR or better per investigator review according to RECIST version 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (8):
- United States (3):
  - NEXT Oncology - San Antonio /ID# 278606, San Antonio, Texas
  - Start Mountain Region /ID# 278609, West Valley City, Utah
  - Next Virginia /ID# 278607, Fairfax, Virginia
- Israel (3):
  - The Chaim Sheba Medical Center /ID# 278416, Ramat Gan, Tel Aviv
  - Rambam Health Care Campus /ID# 278418, Haifa
  - Hadassah Medical Center-Hebrew University /ID# 278420, Jerusalem
- Japan (2):
  - Saitama Medical University International Medical Center /ID# 278437, Hidaka, Saitama
  - Shizuoka Cancer Center /ID# 278538, Sunto-gun, Shizuoka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-760